CLINICAL TRIAL: NCT02742051
Title: A Randomised Pilot Study of Neoadjuvant Everolimus Plus Letrozole Compared With FEC in Postmenopausal Patients With ER-positive, HER2-negative Breast Cancer
Brief Title: A Trial of Neoadjuvant Everolimus Plus Letrozole Versus FEC in Women With ER-positive, HER2-negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jieqiong Liu, M.D., Ph.D., Attending Surgeon of Breast Tumor Center, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 50102016015
Record Dates: First submitted 2016-04-07; First posted 2016-04-18 (Estimated); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus; Letrozole; Fluorouracil; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Everolimus+Letrozole (Experimental): everolimus 10mg/d,po + letrozole 2.5mg/d,po * 18 weeks
  Interventions: Drug: Everolimus; Drug: Letrozole
- Fluorouracil+epirubicin+cyclophosphamide (Active Comparator): Fluorouracil 600mg/m2,iv,d1 + epirubicin 90mg/m2,iv,d1 + cyclophosphamide 600mg/m2,iv,d1 * 6 cycles (every 21 days per cycle)
  Interventions: Drug: Fluorouracil; Drug: Epirubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Everolimus — Neoadjuvant endocrine therapy
  Other Names: RAD001
  Arms: Everolimus+Letrozole
Drug: Letrozole — Neoadjuvant endocrine therapy
  Other Names: Femara
  Arms: Everolimus+Letrozole
Drug: Fluorouracil — Neoadjuvant chemotherapy
  Other Names: 5-Fu
  Arms: Fluorouracil+epirubicin+cyclophosphamide
Drug: Epirubicin — Neoadjuvant chemotherapy
  Other Names: EPB
  Arms: Fluorouracil+epirubicin+cyclophosphamide
Drug: Cyclophosphamide — Neoadjuvant chemotherapy
  Other Names: CTX
  Arms: Fluorouracil+epirubicin+cyclophosphamide

SUMMARY:
This open, randomized pilot feasibility trial is to evaluate the feasibility and effect of neoadjuvant everolimus plus letrozole versus neoadjuvant fluorouracil, epirubicin plus cyclophosphamide (FEC) in treating postmenopausal women with ER-positive, HER2-negative breast cancer. Forty postmenopausal stage M0, ER-positive, HER2-negative invasive breast cancer women who had a primary tumor > 2cm by imaging or an axillary lymph node > 2cm by imaging were randomly (1:1) enrolled to receive neoadjuvant everolimus plus letrozole for 18 weeks or neoadjuvant FEC for 6 cycles before surgery. The primary objective is to determine the feasibility of neoadjuvant everolimus plus letrozole in postmenopausal patients with ER-positive, HER2-negative breast cancer. Secondary aims are to compare the ultrasound response rate, pathological complete response (pCR) rate, breast-conserving surgery rate, toxicities, and changes in the percentages or counts of peripheral blood CD4+ T cells, CD8+ T cells, tumor-specific CTLs, T helper cells (Th), regulatory T cells (Treg), and NK cells and changes in tumor Ki67 index (pre- versus post- neoadjuvant therapy).

ELIGIBILITY:
Inclusion Criteria:

* The patients signed the written informed consent
* The patients present with non-metastatic unilateral invasive ER-positive, HER2-negative breast cancer with a primary breast tumor > 2cm by imaging or an axillary lymph node > 2cm by imaging.
* Postmenopausal women with age less than 70 years old.
* The patients have no history of hormone therapy, chemotherapy, breast cancer surgery and radiotherapy.
* The patients have normal cardiac functions by echocardiography.
* The patients' ECOG scores are ≤2.
* The patients can swallow pills.
* The results of patients' blood tests are as follows:

  * Hb≥90g/L;
  * WBC≥4E+9/L;
  * Plt≥100E+9/L;
  * Neutrophils≥1.5E+9/L;
  * ALT and AST ≤ triple of normal upper limit;
  * TBIL ≤ 1.5 times of normal upper limit;
  * Creatinine ≤ 1.5 times of normal upper limit.

Exclusion Criteria:

* The patients have other cancers at the same time or have the history of other cancers except controlled skin basal cell carcinoma or skin squamous cell carcinoma or carcinoma in situ of cervix uterus;
* The patients have active infections that were not suitable for chemotherapy;
* The patients have severe non-cancerous diseases.
* The patients have bilateral breast cancers or multifocal breast cancers or inflammatory breast cancers.
* The patients have a history of previous treatment with mTOR inhibitors.
* The patients are undergoing current administration of anti-cancer therapies, or are attending other clinical trials.
* The patients are in some special conditions that they cannot understand the written informed consent, such as they are demented or hawkish.
* The patients have allergic history or contraindication of any of the interventional drugs.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-03-14 (Actual); Study Completion 2020-03-14 (Actual)

PRIMARY OUTCOMES:
Feasibility of the trial | during on-neoadjuvant therapy period (defined as the period from the first dose of study medication up to 30 days of the last dose)

SECONDARY OUTCOMES:
Ultrasound response rate | at definitive surgery (18-20 weeks after the first dose of study medication)
Pathological complete response (pCR) rate | at definitive surgery (18-20 weeks after the first dose of study medication)
Breast-conserving surgery rate | at definitive surgery (18-20 weeks after the first dose of study medication)
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | during on-neoadjuvant therapy period (defined as the period from the first dose of study medication up to 30 days of the last dose)
Peripheral blood CD8+ T cell percentage change in relation to neoadjuvant therapy | at definitive surgery (18-20 weeks after the first dose of study medication)
Peripheral blood T helper cell percentage change in relation to neoadjuvant therapy | at definitive surgery (18-20 weeks after the first dose of study medication)
Peripheral blood regulatory T cell percentage change in relation to neoadjuvant therapy | at definitive surgery (18-20 weeks after the first dose of study medication)
Peripheral blood NK cell percentage change in relation to neoadjuvant therapy | at definitive surgery (18-20 weeks after the first dose of study medication)
Blood tumor-specific CTLs count change in relation to neoadjuvant therapy | at definitive surgery (18-20 weeks after the first dose of study medication)
Peripheral blood CD4+ T cell percentage change in relation to neoadjuvant therapy | at definitive surgery (18-20 weeks after the first dose of study medication)
Tumor Ki67 index change in ralation to neoadjuvant therapy | at definitive surgery (18-20 weeks after the first dose of study medication)

CONTACTS AND LOCATIONS:
Overall Officials: Jieqiong Liu, M.D.,Ph.D., Principal Investigator — Breast Tumor Center, Sun Yat-sen Memorial Hospital
Locations (1):
- Sun-Yat-Sen Memorial Hospital of Sun-Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wu W, Chen J, Deng H, Jin L, He Z, Rao N, Nie Y, Yao Y, Yang Y, Su F, Liu J. Neoadjuvant everolimus plus letrozole versus fluorouracil, epirubicin and cyclophosphamide for ER-positive, HER2-negative breast cancer: a randomized pilot trial. BMC Cancer. 2021 Jul 27;21(1):862. doi: 10.1186/s12885-021-08612-y. PMID 34315439
- [Derived] Wu W, Deng H, Rao N, You N, Yang Y, Cao M, Liu J. Neoadjuvant everolimus plus letrozole versus fluorouracil, epirubicin and cyclophosphamide for ER-positive, HER2-negative breast cancer: study protocol for a randomized pilot trial. Trials. 2017 Oct 25;18(1):497. doi: 10.1186/s13063-017-2228-5. PMID 29070044